CLINICAL TRIAL: NCT03423134
Title: A Pilot Evaluation of Newly Developed Adhesives and How They Are Impacted by Out-put
Brief Title: Investigating the Performance of a New Adhesive Strip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_19
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of new adhesive strip (Experimental): A new adhesive strip will be tested in this investigation
  Interventions: Other: New adhesive strip

INTERVENTIONS:
Other: New adhesive strip — This is a strip made of a newly developed adhesive

SUMMARY:
This study investigates the performance of a new adhesive

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had a stoma for more than one year
4. Have intact skin on the area used in the evaluation
5. Has a stoma with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Actively participating in other interventional clinical investigations or have previously participated in this investigation.

5.1. Exception: Participation in other Coloplast in-house clinical investigations are accepted under the circumstances of otherwise complying with the Inclusion and exclusion criteria of this protocol (CP265)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
trans epidermal water loss | 24 hours
  The trans epidermal water loss is a measure for the skins barrier function. There is always a loss of water from the skin due to evaporation. When the skin barrier is damaged the evaporation of water increases. Thus, trans epidermal water loss can be used to assess skin damage

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, Principal Investigator — Head of the pre-clinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark